CLINICAL TRIAL: NCT01776515
Title: A Randomized, Double-blind, Active-controlled, Parallel, Multicenter Phase 3 Study of Tramadol Hydrochloride/Acetaminophen SR Tab. & Tramadol Hydrochloride/Acetaminophen Tab. in Low Back Pain Patients
Brief Title: Phase 3 Study of Tramadol Hydrochloride/Acetaminophen SR Tab. & Tramadol Hydrochloride/Acetaminophen Tab. in Low Back Pain Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW 0919 301 Version 1.00
Record Dates: First submitted 2013-01-21; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; Wontran; Wontran SR Tab.; Tramadol Hydrochloride/Acetaminophen
MeSH Terms: conditions — Low Back Pain | interventions — Tramadol; Acetaminophen

ARMS (2):
- Tramadol hydrochloride/Acetaminophen Tab. (Active Comparator)
  Interventions: Drug: Tramadol hydrochloride/Acetaminophen Tab.
- Tramadol hydrochloride/Acetaminophen SR Tab. (Experimental)
  Interventions: Drug: Tramadol hydrochloride/Acetaminophen SR Tab.

INTERVENTIONS:
Drug: Tramadol hydrochloride/Acetaminophen Tab.
  Arms: Tramadol hydrochloride/Acetaminophen Tab.
Drug: Tramadol hydrochloride/Acetaminophen SR Tab.
  Arms: Tramadol hydrochloride/Acetaminophen SR Tab.

SUMMARY:
The purpose of this study is to evaluate effectness of Tramadol Hydrochloride/Acetaminophen SR Tab. and Tramadol Hydrochloride/Acetaminophen Tab. in patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males/Females aged over 20 years
2. Patient with low back pain who needs analgesic administration
3. Patient with low back pain Who correspond with Class 1, 2 in Quebec Task Force Classification
4. Pain VAS Value over 40 mm
5. Subjects who voluntarily or legal guardian agreed with written consent

Exclusion Criteria:

1. Patients with severe GI tract disorder, liver disease, renal disease, heart disease, hypertension
2. Patients with obvious secondary cause(metastatic cancer, fracture, infectious disease)
3. Patients who had taken back surgery within 24 weeks from the screening point
4. Patients who had taken opioid drug, psychotropic drug within 4 weeks from the screening point
5. Patients who had taken steroid drug(oral, injection) within 4 weeks from the screening point

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Changes in '100 mm pain VAS' value from baseline | 0, 1, 7, 14, 28 day